CLINICAL TRIAL: NCT00797017
Title: Impact of Fentanyl Matrix on Improvement of Pain and Functioning in Spinal Disorder-related Pain: Multicenter, Open Label, Prospective, Observational Study
Brief Title: Study on Impact of Fentanyl Matrix on Improvement of Pain and Functioning in Spinal Disorder-related Pain
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015409
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Low Back Pain
Keywords: Chronic Pain; Fentanyl Matrix; Spinal disorder-related pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 001
  Interventions: Drug: fentanyl
- 002
  Interventions: Drug: fentanyl
- 003
  Interventions: Drug: fentanyl
- 004
  Interventions: Drug: fentanyl
- 005
  Interventions: Drug: fentanyl
- 006
  Interventions: Drug: fentanyl
- 007
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — Infection, starting with 12mcg/h (flexible dose)
  Groups: 005
Drug: fentanyl — (CRPS) Complex Regional Pain Syndrome, starting with 12mcg/h (flexible dose)
  Groups: 004
Drug: fentanyl — Bone Fracture, starting with 12mcg/h (flexible dose)
  Groups: 003
Drug: fentanyl — (FBSS) Failed Back Surgery Syndrome, starting with 12mcg/h (flexible dose)
  Groups: 006
Drug: fentanyl — Other Deformity, starting with 12mcg/h (flexible dose)
  Groups: 007
Drug: fentanyl — (LDK) Lumbar Degenerative Kyphosis, starting with 12mcg/h (flexible dose)
  Groups: 002
Drug: fentanyl — Degenerative Spine Disorder, starting with 12mcg/h (flexible dose)
  Groups: 001

SUMMARY:
The purpose of this observational study is to investigate the impact of fentanyl matrix on improvement of pain and functioning in spinal disorder-related chronic pain.

DETAILED DESCRIPTION:
This study is a prospective, open-label, non-interventional study. The objective of the study is to investigate the impact of fentanyl matrix on improvement of pain and functioning after 8-week treatment of fentanyl matrix in the patients who complained of spinal disorder-related chronic pain in clinical practice according to the investigator's discretion. The primary endpoint is a percent of pain intensity difference between baseline and week 8 of the study. Each patients will evaluate their pain intensity every 28 days during the 8 weeks. The secondary objectives are to observe the change in the following variables after administrating fentanyl matrix; K-ODI (Korean version - Oswestry Disability Index) score, sleep disturbance, disturbance of activities of daily living and disturbance of social activities. In addition, Investigator and patient global assessment, patient preference, CGI-I (Clinical Global Impression - Improvement) and Adverse Events will be investigated. LDK: Lumbar degenerative kyphosis, CRPS: Complex Regional Pain SYndrome, FBSS: Failed Back Surgery Syndrome Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients who complain of spinal disorder-related chronic pain persisting for 3 months or longer
* Patients who can fully observe the overall clinical study requirements including K-ODI completion at the investigator's discretion
* Patients who complain of severe pain (NRS score = 7) because pain was not treated enough with the previous analgesic
* Patients who have never been administered fentanyl matrix over the last one month

Exclusion Criteria:

* Patients with a history of the drug or alcohol abuse in the past or now
* Childbearing women who are pregnant or likely to be pregnant during the study period and male patients who are neither infertile nor willing to refrain from sexual relations but whose partner does not conduct an effective contraception (implant, injections, oral contraceptives, intrauterine device, etc.)
* Patients who are unable to use a transdermal system due to skin disease
* Patients with serious mental disorder
* Patients with history of hypersensitivity to opioid analgesics
* Patients with history of CO2 retention
* Patients who are not eligible for the study participation based on warnings, precautions and contra medications in the package insert of the study drug at the investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had unsatisfactory treatment with previous medication (severe pain: NRS = 7) and no experience with fentanyl matrix will be eligible
Sampling Method: Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity with Numeric Rating Scale | baseline, week 4 and week 8

SECONDARY OUTCOMES:
Impact of activity of daily living and social activities | baseline, week 4 and week 8
Investigator and patient global assessment | baseline, week 4 and week 8
CGI-I (Clinical Global Impression) | baseline, week 4 and week 8
K-ODI (Korean version of Oswestry Disability Index) | baseline, week 4 and week 8
Improvement of sleep disturbance | baseline, week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.